CLINICAL TRIAL: NCT01391468
Title: Beneficial Effect of Probiotics on Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, I-Kuan Wang, China Medical University Hospital, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DMR-99-IRB-308
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2015-08-24 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Probiotics; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): cornstarch
  Interventions: Dietary Supplement: Cornstarch
- Probiotics (Experimental): probiotics
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — intervention group receives probiotics containing 10E9 CFU B. bifidum, B. catenulatum, B. longgim, and L. plantarm in 6 months observations
  Arms: Probiotics
Dietary Supplement: Cornstarch — placebo will be given in 6 months
  Arms: Placebo

SUMMARY:
This is a randomized double blinded placebo control studies are performed in Chronic Kidney Disease (CKD) patients. After informed consent, intervention group receives probiotics containing 109 CFU B. bifidum, B.catenulatum, B. longum, and L.plantarm), while placebo group receives corn starch. In the first year the investigators examine the 60 peritoneal dialysis (PD) patients, in the second year the investigators do the 60 hemodialysis (HD) patients, and in the third year the investigators do the 60 stage 3 and 4 CKD patients. Primary endpoint is cardiovascular event, gastrointestinal symptoms, peritonitis in PD patients, and progression of stage 3 and 4 CKD. Values are compared between the groups by unpaired t test. X2 testis used to compare proportions between the groups. Relative risk and the number needed to treat, both with 95% CI, are used to describe the treatment effect of probiotics. A p value less than 0•05 is regarded as statistically significant.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a global health issue that has a substantial impact on affected individuals. The prognosis of dialysis patients is poor with 30 to 50 percent 5 year survival in nondiabetic patients and 25 percent in diabetics. Cardiovascular disease accounts for approximately half of death of dialysis patients Chronic inflammation, which is widely seen in long-term dialysis patients, is associated with malnutrition, atherosclerosis and an increased mortality risk. Inflammatory markers such as C-reactive protein (CRP),IL-6, Il-18 and TNF-α, are elevated in dialysis and can predict cardiovascular event and all-cause mortality.

Probiotics are microorganisms that have beneficial properties for the host. Three described benefits include suppression of growth or epithelial binding/invasion by pathogenic bacteria, improvement of intestinal barrier function and modulation the immune systems.

Several probiotics preparations induce protective cytokines, including IL-10, and suppress proinflammatory cytokines, such as TNF-α and IL-6. Intestinal microflora is deranged in hemodialysis (HD) patients as an increase in aerobic bacteria such as E. coli and a decrease in anaerobic bacteria such as Bifidobacterium. One study reported that oral administration of ifidobacterium longum in a gastroresistant seamless capsule decreases the the pre-HD serum levels of homocysteine and indoxyl sulfate. Another small-scale study from Japan showed that synbiotics containing lactobacilli and can reduce serum level of p-Cresol in HD patients. High-serum p-cresyl sulfate and indoxyl sulfate levels were associated with renal progression. Serum concentrations of p-cresol are independently associated with overall mortality and cardiovascular disease in HD patients. The aim of the study is 1. to evaluate the difference of intestinal microflora between CKD patients and healthy controls; 2. to evaluate whether the investigators can reduce cardiovascular events in CKD patients, and peritonitis in peritoneal dialysis (PD) patients, retard the progression of stage 3 and 4 CKD patients, and decrease circulating inflammatory markers(CRP, IL-6,IL-18, TNF-α), indoxyl sulfate, p-cresol and homocysteine after probiotics treatment.

Randomized double blinded placebo control studies are performed in CKD patients. After informed consent, intervention group receives probiotics containing 109 CFU B. bifidum, B.catenulatum, B. longum, and L.plantarm), while placebo group receives corn starch. In the first year the investigators examine the 60 PD patients, in the second year the investigators do the 60 HD patients,and in the third year the investigators do the 60 stage 3 and 4 CKD patients. Primary endpoint is cardiovascular event, gastrointestinal symptoms, peritonitis in PD patients, and progression of stage 3 and 4 CKD. Values are compared between the groups by unpaired t test. X2 testis used to compare proportions between the groups. Relative risk and the number needed to treat, both with 95% CI, are used to describe the treatment effect of probiotics. A p value less than 0·05 is regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. receiving peritoneal dialysis for more than 3 months, at least 18 years of age, and GFR < 15 ml/min.
2. receiving hemodialysis dialysis for more than 3 months, at least 18 years of age, and GFR < 15 ml/min.
3. Stage 3 and 4 CKD patients

Exclusion Criteria:

* active infectious conditions within the last 30 days,
* pregnancy for female,
* autoimmune disease e.g. SLE.,
* cardiovascular events before.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: I-Kuan Wang, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Probiotics
Started | 24 | 23
Completed | 18 | 21
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Probiotics | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 23 | 47
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  Taiwan | 24 | 23 | 47
IL-6 [Mean (Standard Deviation); unit: pg/ml] — inflammatory cytokine
  pg/ml | 5.27 (12.78) | 6.55 (10.72) | 5.90 (11.71)

OUTCOME MEASURES:

1. Primary Outcome: the Occurrence of Cardiovascular Event and Peritonitis Events
Time Frame: 6 month follow-up
Measure: Number; unit: participants
Arm/Group | Placebo | Probiotics
Number analyzed (Participants) | 18 | 21
participants
  Cardiovascular event | 0 | 0
  Peritonitis event | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Probiotics; Test type: Superiority or Other; p > 0.05, Chi-squared

2. Secondary Outcome: Change of Gastrointestinal Symptoms at 6 Months
Description: The change in gastrointestinal symptom rating scale (min and maximum scores 0-45) after treatment. The total score is reported. The higher scale represents a worse outcome.
Time Frame: 6 months follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Probiotics
Number analyzed (Participants) | 18 | 21
units on a scale | -2.82 (5) | -1.38 (3.25)
Statistical Analysis 1: Comparison: Placebo vs Probiotics; Test type: Superiority or Other; p = 0.744, Wilcoxon (Mann-Whitney)

3. Post Hoc Outcome: Change of Serum Endotoxin Level at 6 Months
Description: endotoxin is a marker of inflammation in chronic kidney disease patients
Time Frame: 6 months follow-up
Measure: Mean (Standard Deviation); unit: EU/ml
Groups:
- Placebo: Placeo group received maltodextrin for 6 months
Arm/Group | Probiotics | Placebo
Number analyzed (Participants) | 21 | 18
EU/ml | -1.31 (1.61) | 0.84 (2.27)
Statistical Analysis 1: Comparison: Probiotics; Test type: Superiority or Other; p = 0.0042, Wilcoxon (Mann-Whitney) — Only the probiotics group arrived at the reported p-value after 6 months

4. Post Hoc Outcome: Change of Serum IL-10 Level at 6 Months
Description: IL-10 is an anti-inflammatory cytokine; The change of serum IL-10 level at 6 months was measured
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Placebo: Plabeco group received maltodextrin for 6 months
Arm/Group | Probiotics | Placebo
Number analyzed (Participants) | 21 | 18
pg/ml | 3.3 (6.37) | -2.09 (6.73)
Statistical Analysis 1: Comparison: Probiotics; Test type: Superiority or Other; p = 0.0099, Wilcoxon (Mann-Whitney) — Only the probiotics group arrived at the reported p-value after 6 months

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Probiotics | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No